CLINICAL TRIAL: NCT04114591
Title: Contributing Factors to Anterior Resection Syndrome and Its Impact on Quality of Life: A Retrospective Cohort Study
Status: Completed | Type: Observational
Sponsor: University of Malta (Other)
Responsible Party: Principal Investigator, Svetlana Doris Brincat, Surgical trainee, University of Malta
Other Study IDs: S07/18
Record Dates: First submitted 2019-09-25; First posted 2019-10-03 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Low Anterior Resection Syndrome; Cancer; Quality of Life
MeSH Terms: conditions — Low Anterior Resection Syndrome; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LARS symptoms: Patient suffering from LARS as identified through LARS questionnaire
  Interventions: Procedure: anterior resection
- No LARS symptoms: Absence of LARS symptoms
  Interventions: Procedure: anterior resection

INTERVENTIONS:
Procedure: anterior resection — The distance from anal verge, preoperative radiotherapy and presence of stoma were analysed
  Other Names: radiotherapy +/- chemotherapy

SUMMARY:
This study adds to the understanding of the contributing factors leading to LARS, the long term effects of this syndrome post-operatively and its impact on quality of life.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients >18 years, under the care of all surgical firms at Mater Dei Hospital, who had undergone anterior resection for rectal cancer between January 2014 and December 2016

Exclusion Criteria:

* colorectal cancer (>15cm) from anal verge
* permanent stoma
* known disseminated or recurrent disease,
* patient without restitution of bowel continuity after 1 year

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult patients >18 years, under the care of all surgical firms at Mater Dei Hospital, who had undergone anterior resection for rectal cancer between January 2014 and December 2016
Sampling Method: Non-Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
LARS incidence | 1 year
  Incidence of LARS in patients who had anterior resection
Risk factors | 1 year
  Variable factors which might have contributed to LARS were the following:
  * Age
  * Gender
  * Diabetes mellitus
  * Pathological stage
  * MRI stage
  * Distance from anal verge
  * Surgical technique
  * Preoperative radiotherapy
  * Preoperative chemotherapy
  * Postoperative radio/chemotherapy
  * Type of anastomosis
  * Presence of stoma
  * Interval from stoma reversal
  * Duration of follow-up
Life | 1 year
  The association between LARS and quality of life was assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Svetlana Doris Brincat, Principal Investigator — Mater Dei Hospital
Locations (1):
- Mater Dei Hospital, Valletta, Malta

IPD SHARING:
Plan to Share IPD: Undecided